CLINICAL TRIAL: NCT01623336
Title: Safety and Efficacy of BIP48 (Peginterferon Alfa 2b 48kDa) Compared With Pegasys® (Peginterferon 2a 40kDa) for Treatment of Chronic Hepatitis C: Randomized, Multicentric Study With Blinded Analysis
Brief Title: BIP48 (Peginterferon Alfa 2b 48kDa) Compared With Pegasys® (Peginterferon 2a 40kDa) for Treatment of Chronic Hepatitis C
Acronym: BIP48II/III
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/0468
Record Dates: First submitted 2012-06-13; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Hepatitis C
Keywords: HEPATITIS; HEPATITIS C; PEGINTERFERON; BIOEQUIVALENCE; TREATMENT
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis; Hepatitis C | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pegasys ® (Active Comparator): Patients will receive Pegasys ® (peginterferon alfa-2a 40kDa) at a dose of 180 micrograms, subcutaneously, once a week, associated with ribavirin at a dose 1000-1250 mg,daily. For genotype 1 treatment time is 48 to 72 weeks and for genotypes 2 and 3, 24 weeks.
  Interventions: Drug: BIP 48 (Peginterferon alfa 2b 48kDA); Drug: Peginterferon alfa 2a 40kDA
- BIP 48 (Peginterferon alfa 2b 48kDA) (Experimental): Patients will receive BIP 48, 180 micrograms a week, SC, for the same period as Pegasys ®.
  Interventions: Drug: BIP 48 (Peginterferon alfa 2b 48kDA)

INTERVENTIONS:
Drug: BIP 48 (Peginterferon alfa 2b 48kDA) — BIP 48 (Peginterferon alfa 2b 48kDA)will be administered in a dose of 180 micrograms, once a week, subcutaneous, for 24 to 48 weeks to genotypes 2 and 3, and for 48 to 72 weeks to genotype 1.
  Arms: Pegasys ®
Drug: Peginterferon alfa 2a 40kDA — Patients will receive Pegasys ® in a dosage of 180 micrograms, once a week, subcutaneous, for 24 to 48 weeks to genotypes 2 and 3 and for 48 to 72 weeks to genotype 1.
  Other Names: Pegasys ®
  Arms: Pegasys ®
Drug: BIP 48 (Peginterferon alfa 2b 48kDA) — Patients will receive BIP 48 in a dosage of 180 micrograms, once a week, subcutaneous, for 24 to 48 weeks to genotypes 2 and 3 and for 48 to 72 weeks to genotype 1.
  Arms: BIP 48 (Peginterferon alfa 2b 48kDA)

SUMMARY:
The purpose of the study is to demonstrate the noninferiority of BIP48 (48 kDa peginterferon alfa-2b) compared to Pegasys ® (40 kDa peginterferon alfa-2a) associated with ribavirin, in naive patients with chronic hepatitis C.

DETAILED DESCRIPTION:
The study will be an open, multicenter, randomized, controlled phase II - III trial. Patients (n = 740) will be randomized (1:1) to receive BIP48 (peginterferon alfa-2b 48kDa) or Pegasys ® (peginterferon alfa-2a 40kDa) 180 micrograms ,subcutaneously,once a week,associated with ribavirin at a dose 1000-1250 mg, orally, daily. For genotype 1 treatment time will be 48 to 72 weeks and for genotypes 2 and 3, 24 to 48 weeks. The study's population will be naive patients, of both sex, between 18 and 70 years old, with chronic hepatitis C (HCV), genotypes 1, 2 or 3, from 18 to 25 Brazilian research centers. Diagnostic criteria will be as followed: positive anti-HCV and qualitative PCR, liver biopsy showing any degree of fibrosis and at least mild inflammatory activity, performed in the last 24 months. The interruption Criteria will be: no partial virological response at 12 weeks and positive quantitative PCR at week 24.The primary outcome will be the rate of sustained virologic response and the secondary endpoints will be the quality of life during treatment, frequency of adverse events and cost-effectiveness. As a substudy, will be performed a comparative assessment in 24 patients, evaluating viral kinetics, pharmacokinetics and pharmacodynamics of repeated doses of both alfapeginterferons .

ELIGIBILITY:
Inclusion Criteria:

1. anti-HCV positive;
2. viral load of HCV positive;
3. viral genotypes 1, 2 or 3;
4. the absence of previous treatment for chronic hepatitis C;
5. liver biopsy performed in the last 36 months classified by Metavir score as at least A1, with any degree of fibrosis ;
6. age from 18 to 70 years old;
7. hemoglobin greater than 11 g / dl;
8. platelet count higher than 75.000/mm3;
9. neutrophils higher than 1.500/mm3;
10. use of, at least two contraceptive methods during treatment and up to 36 weeks after the last dose of study medication (for male or female subjects in fertile age );
11. concordance and signing of the informed consent.

Exclusion Criteria:

1. decompensated cirrhosis (Child-Pugh score> 6);
2. history of bleeding gastroesophageal varices;
3. hemoglobinopathies;
4. hepatocellular carcinoma;
5. co-infection with HIV or HBV;
6. other coexisting chronic liver disease, as autoimmune hepatitis, Wilson disease, hemochromatosis, chronic obstructive cholestatic disease or autoimmune disease, alcoholic liver disease;
7. malignancies except basal cell carcinoma in situ or cervix carcinoma;
8. systemic autoimmune diseases, except compensated autoimmune thyroid diseases ;
9. uncontrolled seizures;
10. primary immunodeficiencies;
11. myelosuppression;
12. coagulation disorders;
13. thrombophilias;
14. thrombopathy ;
15. decompensated heart failure;
16. chronic renal failure;
17. diagnosis of other comorbidity that would compromise the subject's participation in the research study as judged by the investigator (eg, neuropsychiatric diseases, systemic infection or antibiotic use within 4 weeks, decompensated diabetes mellitus, ischemic heart disease, heart failure, respiratory or renal or uncontrolled hypertension);
18. prior organ transplantation, except cornea;
19. alcohol consumption exceeding 20g/day for women and 40g/dia for men during the past six months;
20. use of illicit drugs in the previous six months;
21. use of immunosuppressive agents during the previous six months;
22. pregnancy or lactation;
23. male research subjects whose sexual partner is pregnant;
24. previous treatment with IFN or ribavirin in the last 6 months prior to inclusion;
25. subjects with hypersensibility to IFN alpha and / or any of its components;
26. subjects with hypersensibility to ribavirin and / or any of its ingredients;
27. participation in another clinical study in the last 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The rate of sustained virologic response - SVR - measured by PCR at 24 weeks after treatment. | HCV PCR will be measured at 24 weeks after the end of therapy (week 48 for genotypes 2 and 3 and week 72 for genotype 1)

SECONDARY OUTCOMES:
Frequency of adverse events | Clinical exam, blood tests and immunogenicity evaluation will be done twice monthly, in the first month, and then monthly until the end of treatment( week 24 for genotypes 2 and 3 and week 48 for genotype 1).
  Blood tests included: ALT, AST, Creatinine and complete blood count. Anti-interferon immunoglobulin and thyroid-stimulating hormone (TSH) will be measured in the weeks 12, 24, 36, 48, 60 and 72 of the study.
Virologic response at the end of treatment | Viral load will be measured at the end of treatment (week 24 for genotypes 2 and 3 and week 48 for genotype 1)
  Viral load will be measured by quantitative PCR at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo D. Picon, Invest, Principal Investigator — Hospital de Clínicas de Porto Alegre; Guilherme B. Sander, Coord, Study Director — Hospital de Clínicas de Porto Alegre; Luiz E. Mazzoleni, Coord, Study Director — Hospital de Clínicas de Porto Alegre; André C. Wortmann, Monitor, Study Chair — NUCLIMED; Karine M. Amaral, Coordenação, Study Chair — NUCLIMED; Marisa B. Costa, Sub Coord, Study Chair — NUCLIMED; Tobias C. Milbradt, Coord Log., Study Chair — NUCLIMED; Indara C. Saccilotto, Coordenação, Study Chair — NUCLIMED; Amanda Quevedo, Sub Coord, Study Chair — NUCLIMED; Daiana V. Gomes, AssitSocial, Study Chair — NUCLIMED
Locations (1):
- Ufrgs/Hcpa, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] da Silva AMV, Alvarado-Arnez LE, Azamor T, Batista-Silva LR, Leal-Calvo T, Bezerra OCL, Ribeiro-Alves M, Kehdy FSG, Neves PCDC, Bayma C, da Silva J, de Souza AF, Muller M, de Andrade EF, Andrade ACM, Dos Santos EM, Xavier JR, Maia MLS, Meireles RP, Cuni HN, Sander GB, Picon PD, Matos DCS, Moraes MO. Interferon-lambda 3 and 4 Polymorphisms Increase Sustained Virological Responses and Regulate Innate Immunity in Antiviral Therapy With Pegylated Interferon-Alpha. Front Cell Infect Microbiol. 2021 Jul 7;11:656393. doi: 10.3389/fcimb.2021.656393. eCollection 2021. PMID 34307188